CLINICAL TRIAL: NCT04774627
Title: Pancytopenia Related to PARP Inhibitors in Cancer Patients : an Observational and Retrospective Study Using the WHO's Pharmacovigilance Database (PancytoRIB)
Brief Title: Pancytopenia Related to PARP Inhibitors (PancytoRIB)
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: Pharmaco 20200210
Record Dates: First submitted 2021-02-25; First posted 2021-03-01 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-02

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Poly(ADP-ribose) Polymerase Inhibitors; olaparib; rucaparib; niraparib; talazoparib; veliparib; pamiparib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: PARP inhibitor — All patients treated at least with 1 PARPi
  Other Names: olaparib, rucaparib, niraparib, talazoparib, veliparib, pamiparib

SUMMARY:
Although PARP inhibitors (PARPi) have proved effective in treating many cancers, few patients receiving PARPi may experience rare but serious adverse events such as pancytopenia. Today, data about pancytopenia are scarce.

The objective was to investigate reports of pancytopenia adverse events related to PARPi, including olaparib, rucaparib, niraparib, talazoparib, veliparib and pamiparib using the World Health Organization's (WHO) pharmacovigilance database: VigiBase.

DETAILED DESCRIPTION:
Here, investigators use the World Health Organization's (WHO) database of individual safety case reports, to identify cases of pancytopenia related to PARPi.

ELIGIBILITY:
Inclusion Criteria:

* case reported in the World Health Organization (WHO) database (VigiBase) of individual safety case reports at the time of the extraction,
* patients treated with at least 1 PARPi (with ATC classification system): olaparib (ATC L01XX46), niraparib (ATC L01XX54), rucaparib (ATC L01XX55), talazoparib (ATC L01XX60), veliparib (none) and pamiparib (none).

Exclusion Criteria: chronology not compatible between the PARPi and adverse event.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cancer patients treated with PARPi and experiencing pancytopenia.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-02-07 (Actual); Primary Completion 2021-02-27 (Actual); Study Completion 2021-03-24 (Actual)

PRIMARY OUTCOMES:
Pancytopenia reports related to PARPi. | From inception to Feb, 2021
  Identification of the pancytopenia adverse event related to PARP inhibitors reported in the World Health Organization's (WHO) database of individual safety case reports.

SECONDARY OUTCOMES:
Description of the latency period since first PARPi exposure. | From inception to Feb, 2021
Description of the fatality rate. | From inception to Feb, 2021
Description of patients who experienced co-reported adverse events | From inception to Feb, 2021

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandre Joachim, Caen, Basse Normandie, France